CLINICAL TRIAL: NCT05445882
Title: A Phase II Study of N-803 Alone or in Combination With BN-Brachyury Vaccine or Bintrafusp Alfa (M7824) for Participants With Castration Resistant Prostate Cancer
Brief Title: N-803 Alone or in Combination With BN-Brachyury Vaccine or Bintrafusp Alfa (M7824) for Participants With Castration Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed by study team, no subjects enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000309; 000309-C
Record Dates: First submitted 2022-07-02; First posted 2022-07-06 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2021-04

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: Pd-L1 Inhibitor; Il-15/ Il-15ra; Tgf-SS- Trap; Crpc
MeSH Terms: interventions — bintrafusp alfa protein, human; ALT-803

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): N-803 + BN-Brachyury (+ bintrafusp alfa if progression beyond 12 weeks)
  Interventions: Drug: N-803; Biological: BN-Brachyury
- Arm 2 (Experimental): N-803 (+ BN-Brachyury + bintrafusp alfa if progression beyond 12 weeks)
  Interventions: Drug: N-803
- Arm 3 (Experimental): N-803 + bintrafusp alfa (+ BN-Brachyury if progression beyond 12 weeks)
  Interventions: Drug: Bintrafusp alfa; Drug: N-803

INTERVENTIONS:
Drug: Bintrafusp alfa — Bintrafusp alfa (1,200 mg) will be given via IV infusion every 2 weeks for up to 3 years.
  Arms: Arm 3
Drug: N-803 — N-803 (15 mcg/kg) subcutaneous injection will be given every 2 weeks for up to 3 years.
Biological: BN-Brachyury — BN-Brachyury collectively refers to the priming doses (MVA-BN-Brachyury) and the boost doses (FPV-Brachyury). MVA-BN-Brachyury subcutaneous injection will be given as 2 priming doses 2 weeks apart. FPV-Brachyury subcutaneous injection will follow MVA-BN-Brachyury injection 2 weeks later every month for 6 months total, then every 3 months until reaching 2 years. After 2 years FPV-Brachyury may be continued at 6-month dosing intervals for up to 3 years.
  Arms: Arm 1

SUMMARY:
Background:

Prostate cancer does not trigger a strong immune response in the body. Hormone therapy, to reduce levels of testosterone in the body, can be helpful to treat some prostate cancers. However, castration-resistant prostate cancer (CRPC) keeps growing even when the testosterone is reduced to a very low level. Men with metastatic CRPC survive an average of only 3 years. More effective treatments are needed.

Objective:

To test whether an immunotherapy drug (N-803), alone or in combination with other drugs, can help treat CRPC.

Eligibility:

Males aged 18 or older with CRPC. Prior treatment with testosterone-lowering therapy is required.

Design:

Participants will be screened. They will have blood and urine tests. They will have a CT scan of the chest, abdomen, and pelvis.

They will continue to receive hormone therapy for prostate cancer.

Participants will come to the NIH clinic once a week for the first 4 weeks. Then they will come once every 2 weeks. Visits will last up to 8 hours. The study will continue up to 3 years.

All participants will receive N-803 once every 2 weeks. The drug is injected just under the skin with a small needle.

Some participants will receive N-803 plus another drug (brachyury vaccine). This drug is also injected under the skin with a small needle.

Some participants will receive N-803 plus a different drug (bintrafusp alfa) once every 2 weeks. This drug is given through a tube attached to a needle placed in a vein in the arm.

Some participants may receive all 3 drugs.

Participants will have imaging scans every 12 weeks.

DETAILED DESCRIPTION:
BACKGROUND:

* Prostate cancer is poorly recognized by T cells. Lack of an immune response is one explanation for the lower response rates (<15%) observed with anti-PD-1/PD-L1 therapies for prostate cancer.
* BN-Brachyury is a novel recombinant vector-based therapeutic cancer vaccine designed to induce an enhanced immune response against brachyury, which is overexpressed in many solid tumor types, including prostate adenocarcinoma. BN-Brachyury collectively refers to the priming doses (MVA-BN-Brachyury) and the boost doses (FPV-Brachyury) of the vaccine platform.
* Bintrafusp alfa is a bifunctional fusion protein consisting of an anti-programmed death ligand 1 (PD-L1) antibody and the extracellular domain of transforming growth factor beta (TGF-beta) receptor type 2, a TGF-beta trap. Bintrafusp alfa can also mediate antibody-dependent cellular cytotoxicity in vitro.
* N-803 is an IL-15/IL-15Ralpha superagonist complex that can enhance natural killer (NK) cell-mediated antibody-dependent cellular cytotoxicity (ADCC) and T-cell cytotoxicity.
* Synergistic anti-tumor effects have been observed in vitro when combining bintrafusp alfa and N-803, and in vivo when combining these agents with tumor vaccine in animal models.
* Given the high response rate of 46% seen thus far with the combination of BN-Brachyury, bintrafusp alfa, and N-803 in Arm 2.2A of QuEST1 trial suggests that it is important to determine the relative contribution of each agent in order to determine if a subset of these agents can be used while preserving efficacy and minimizing toxicity. In particular, because the combination of bintrafusp alfa with BN-Brachyury did not produce a significant response rate until N-803 was added, the objective of this Confirmatory QuEST1 trial (ConQuEST) is to investigate the impact of N-803 alone or in an unstudied combination with either BN-Brachyury or bintrafusp alfa.
* This trial offers a means to enhance response rates in castration-resistant prostate cancer (CRPC) on a potentially shorter timeline than with that of traditional trial designs.

OBJECTIVE:

-To determine the clinical efficacy of N-803 alone or in combination with brachyury vaccine or bintrafusp alfa among participants with CRPC

ELIGIBILITY:

* Participants must have castration-resistant prostate cancer. Prior treatment with testosterone lowering therapy for CRPC is required.
* Castrate testosterone level (<50 ng/dl or 1.7nmol /L)
* Age >=18 years
* ECOG performance status <=1

DESIGN:

* This is an open label, non-randomized, Phase II trial with sequential enrollment into Arm 1 followed by Arms 2 or 3 depending on the response to treatment.
* Enrollment will begin with Arm 1 (N-803 + brachyury vaccine), and response will be defined as objective response by response evaluation criteria in solid tumors (RECIST) 1.1 criteria or sustained prostate-specific antigen (PSA) decrease >= 30% for > 21 days.
* If at least 3 responses out of 12 participants are seen in Arm 1 within the first 12 weeks of treatment initiation, enrollment will begin with Arm 2 (N-803 alone); whereas, if fewer than 3 responses out of 12 participants, enrollment will begin in Arm 3 (N-803 + bintrafusp alfa).
* Bintrafusp alfa (1,200 mg) will be given via IV infusion every 2 weeks.
* N-803 (15 mcg/kg) subcutaneous injection will be given every 2 weeks.
* MVA-BN-Brachyury subcutaneous injection will be given as 2 priming doses 2 weeks apart. Each dose will comprise 4 x 0.5 mL subcutaneous injections consisting of a nominal virus titer of 2.0 x 10^8 infectious units (Inf.U).
* FPV-Brachyury subcutaneous injection will follow MVA-BN-Brachyury injection 2 weeks later every month for 6 months total, then every 3 months until reaching 2 years. After 2 years FPV-Brachyury may be continued at 6-month dosing intervals. Each dose will be a 0.5 mL injection consisting of a nominal virus titer of 1 x 10^9 Inf.U.
* Participants who respond or have the stable disease will continue on their assigned treatment regimen with the possibility of switching to triplet therapy (N-803 + brachyury vaccine + bintrafusp alfa) on PSA or radiographic progression if clinically stable should they experience progression beyond 12 weeks. Anyone who progresses clinically at any point during treatment will be taken off treatment, and anyone who progresses radiographically on triplet therapy will be taken off treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:
* History of castration-resistant prostate cancer (CRPC) with histologic confirmation of diagnosis at any time point prior to initiation of study therapy. Note: If a pathology report is unavailable, a history consistent with prostate cancer is sufficient.
* Prior treatment with testosterone lowering therapy for CRPC is required.
* Castrate testosterone level (<50ng/dl or 1.7nmol /L).
* Radiological confirmation of metastatic disease

OR

-Progressive disease at study entry defined as one or more of the following criteria occurring in the setting of castrate levels of testosterone:

--radiographic progression defined as any new or enlarging bone lesions or growing lymph node disease, consistent with prostate cancer

OR

* PSA progression defined by sequence of rising values separated by >1 week (2 separate increasing values over a minimum of 1 ng/ml (Prostate Cancer Working Group 3 (PCWG3) PSA eligibility criteria). If participants had been on flutamide, PSA progression is documented 4 weeks or more after withdrawal. For participants on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal. The requirement for a 4-6-week withdrawal period following discontinuation of flutamide, nilutamide, or bicalutamide only applies to participants who have been on these drugs for at least the prior 6 months. For all other participants, they must stop bicalutamide, nilutamide, or flutamide prior to treatment initiation.

  * Participants are willing to continue androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone analog/antagonist or bilateral orchiectomy.
  * Age >=18 years.
  * ECOG performance status <= 1
  * Participants must have adequate organ and marrow function as defined below:
* Absolute neutrophil count >= 1000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin within normal institutional limits; in participants with Gilbert s, <= 3.0 mg/dL
* AST (SGOT)/ALT (SGPT) <= 2.5X upper limit of normal. For subjects with liver involvement in their tumor, AST <= 3.5 (SqrRoot) ULN, ALT <= 3.5 (SqrRoot) ULN, and bilirubin <= 3.0 is acceptable
* Creatinine within 1.5X upper limit of normal institutional limits

  * Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry, during the study, and maintain such contraception until 4 months following the last dose of any study agent.
  * Human immunodeficiency virus (HIV)-positive participants must have CD4 count >= 200 cells per cubic millimeter before treatment initiation, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman s disease

within 12 months prior to treatment initiation.

* Participants with successfully treated HCV if HCV viral load is undetectable.
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Participants who are immunocompromised as follows:

  * Chronic administration (defined as daily or every other day for continued use >14 days) of systemic corticosteroids or other immune suppressive drugs, within 28 days before treatment initiation. NOTE: Systemic corticosteroids at physiologic doses <= 10 mg/day of prednisone or equivalent and steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed. Nasal, or inhaled steroid, topical steroid creams, and eye drops for small body areas are also allowed.
  * History of allogeneic peripheral stem cell transplantation, or solid organ transplantation requiring immunosuppression.
* Active autoimmune disease, except: participants with type 1 diabetes mellitus, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring current immunosuppression, or with other endocrine disorders on replacement hormones if the condition is well controlled.
* History of prostate cancer with brain/leptomeningeal metastasis. Note: Except if status post definitive radiotherapy or surgery and are asymptomatic.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents to be used.
* Known allergy to eggs, egg products, aminoglycoside antibiotics (e.g., gentamicin or tobramycin).
* Prior investigational drug, chemotherapy, immunotherapy, or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to treatment initiation. Note: except if all treatment-related toxicities have resolved or are minimal and the participant meets all other eligibility criteria.
* Participants who have had cytotoxic chemotherapy for metastatic castration-resistant prostate cancer within the past year. NOTE: Participants who have had docetaxel for metastatic castration sensitive prostate cancer per CHAARTED data may enroll as long as they did not have progressive disease while on docetaxel and are 3 months removed from treatment, with all treatment-related toxicities resolving to at least grade 1.
* Uncontrolled intercurrent acute or chronic illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (>New York Heart Association Class I), hepatic disease, unstable angina pectoris, serious cardiac arrhythmia, requiring medication, uncontrolled hypertension (SBP>170/ DBP>105) or psychiatric illness/social situations within 12 months before treatment initiation that would limit compliance with study requirements.
* History of bleeding diathesis or recent major bleeding events (i.e. Grade >= 2 bleeding events within 4 weeks prior to study treatment initiation)
* Subjects unwilling to accept blood products or blood transfusions as medically indicated. As there is a risk of severe bleeding with M7824, participants must be willing to receive blood transfusions if medically necessary for their own safety
* Subjects who received a live vaccine within 4 weeks or COVID-19 vaccines within 2 weeks prior to the study treatment initiation.
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto).
* Major surgery within 4 weeks before treatment initiation. NOTE: A biopsy will not preclude a subject from starting the study.
* History of hepatitis B (HBV) infection.
* Use of regularly scheduled opiate analgesics for prostate cancer-related pain.
* Subjects unwilling to accept blood products as medically indicated
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial (including the long-term follow-up), or would interfere with the evaluation of the trial endpoints.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy of N-803 alone or in combination with brachyury vaccine or bintrafusp alfa | 12 weeks
  In each arm, the fraction who experience a response by 12 weeks will be noted and reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Duration of response | 3 years
  the date of response until the date of progression or other determination that the response has ended
Radiographic response | 3 years
  The fraction of participants with a radiographic response will be noted along with a 95% confidence interval, separately for each arm based on imaging
Safety profile of N-803 alone or in combination with brachyury vaccine or bintrafusp alfa | 3 years
  the number of participants with toxicities experienced by grade and type, by arm, as well as overall.

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000309-C.html